CLINICAL TRIAL: NCT01338298
Title: Double-Blind Placebo Controlled Study of Adjunctive Aripiprazole for Symptomatic Hyperprolactinemia In Premenopausal Women With Schizophrenia
Acronym: DAAMSEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, MPRC, Deanna L. Kelly, Pharm.D., BCPP, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00047496, HP-00055154
Record Dates: First submitted 2011-04-17; First posted 2011-04-19 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Hyperprolactinemia
Keywords: Schizophrenia; Symptomatic Hyperprolactinemia; Hormone; Menstrual
MeSH Terms: conditions — Hyperprolactinemia; Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole (Active Comparator)
  Interventions: Drug: Aripiprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole dosing will begin at 5 mg/day once daily and increased to 10mg by mouth once daily at the end of week 2 and then increased to 15 mg/day once daily at the end of week 8 in women who have not yet regained their menstrual period. If a woman gets her menstrual period on the 5 or 10 mg dose she will remain on this dose for the study.
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Placebo — The placebo will be sucrose filled capsules that are identical to the active medication. It is double blind so no one will know if the capsule is placebo or aripiprazole.
  Arms: Placebo

SUMMARY:
Prolactin is a hormone that naturally occurs in the body. Some women taking antipsychotic medications may have high levels of prolactin in their bodies. High levels of prolactin may cause women to have problems with sex or satisfaction from sex. It may also cause women to have fewer or no menstrual periods. It may also cause the production of breast milk and may contribute to long term bone loss.

In this study, the investigators are testing whether taking adding a low dose of an antipsychotic medication called aripiprazole may help improve high prolactin levels and help with sexual dysfunction or problems with menstrual periods. The investigators are also looking to see if it may slow the loss of bones. This medication has been shown to be helpful for improving symptoms of schizophrenia.

DETAILED DESCRIPTION:
This will be a 16-week, double blind, placebo controlled randomized trial of aripiprazole added to an existing stabilized regimen of antipsychotics (either risperidone or paliperidone oral or long acting injectable formulations) for treatment of elevated symptomatic prolactin levels. Aripiprazole dosing will begin at 5 mg/day once daily and increased to 10mg by mouth once daily at the end of week 2 and then increased to 15 mg/day once daily at the end of week 8 in women who have not yet regained their menstrual period. If a woman gets her menstrual period on the 5 or 10 mg dose she will remain on this dose for the study. Women will remain on their current stabilized medication regimen during the course of the adjunctive trial of aripiprazole or placebo. Subjects will be able to receive anticholinergic medications as needed (e.g., benztropine and diphenhydramine) for extrapyramidal side effects, propranolol for akathisia, and benzodiazepines (e.g.,lorazepam) for agitation or anxiety.

Participants will be assigned to either get aripiprazole or placebo (a sugar pill), this will be decided randomly with a 50-50 chance of receiving one or the other medication. The placebo will be sucrose filled capsules that are identical to the active medication. It is double blind so no one will know if the capsule is placebo or aripiprazole. The dosing will be the exact same, one capsule taken daily until week 8. At this time 2 capsules will be given if the participant dose not regains their menstrual period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be females of any race, with an age range of 18?50.
* Subjects will meet DSM-IV TR (APA, 2000) criteria for either schizophrenia, schizoaffective disorder, or bipolar disorder. A best estimate diagnostic approach will be utilized in which information from the Structured Clinical Interview for DSM-IV (First et al, 1997) is supplemented by information from family informants, previous psychiatrists, and medical records to generate a diagnosis
* Women will need to be taking a stable dose of antipsychotic regimen for at least two months and are considered to have stable symptoms by the treating psychiatrist. This regimen must include any form of risperidone or paliperidone.
* All women will have a prolactin level > 24 ng/ml (either identified at screening or from the past 6 weeks in the medical record)
* All women will have evidence of a prolactin related hormonal side effect (amenorrhea, oligomenorrhea or galactorrhea). This will be determined by patient report/history and medical record/clinician interview. Oligomenorrhea is defined as infrequent, irregularly timed episodic bleeding occurring at intervals of more than 35 days from the previous menstrual cycle and amenorrhea is defined as absence of menstruation for three menstrual cycles or 6 months (Berek et al. 2002). Galactorrhea is defined as lactation or copious milk secretion.
* Subjects must be judged competent to participate in the informed consent process and provide voluntary informed consent, by scoring a 10 out of 12 on the Evaluation to Sign Consent (ESC)

Exclusion Criteria:

* Postmenopausal women will be excluded. Since it may be difficult to determine menopause in patients with amenorrhea, any women more than 45 years will be assessed for menopausal symptoms such as but not limited to or by: hot flushes, depression, excitability and fatigue. A medical doctor will advise on the menopausal status.
* Patients with a history of a pituitary tumor (microadenoma, macroadenoma, neoplasm) will not be included in the study. Previous medical records will be obtained if possible to examine prolactin levels and medical histories.
* Subjects with documented Cushing's disease, or who are pregnant or currently lactating post pregnancy will be excluded.
* Subjects who meet DSM-IV TR criteria for alcohol or substance abuse within the last month are excluded. Subjects with nicotine use or dependence will not be excluded.
* Medications which may increase prolactin or cause sexual dysfunction, including: metoclopramide, methyldopa, reserpine, amoxapine, droperidol, prochlorperazine, promethazine, bromocriptine, cabergoline, pergolide, There are many medications that may affect sexual function (not hormonal side effects) unrelated to dopamine transmission. These are only permitted as long as the subject has been receiving them for greater than 4 weeks (SSRIs, mood stabilizers, diuretics, antihypertensives, H2antagonists, bupropion). We allow these medications to enhance generalizability

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, Pharm.D., BCPP, Principal Investigator — University of Maryland, College Park
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aripiprazole | Placebo
Started | 24 | 18
Completed | 20 | 15
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Abdominal Pain and scheduled surgery | 0 | 1
Not completed — Administrative error | 0 | 1
Not completed — Positive symptom worsening | 1 | 0
Not completed — Depressive symptoms and nausea | 1 | 0
Not completed — Non-adherence | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 24 | 18 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 18 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (8.9) | 36.0 (10.1) | 36.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 42
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 18 | 42

OUTCOME MEASURES:

1. Primary Outcome: To Determine if Adjunct Aripiprazole Will Resolve or Improve Prolactin Related Hormonal Side Effects (Amenorrhea, Oligomenorrhea, Galactorrhea).
Description: We will assess this outcome by monitoring the return of menstruation and the elimination of lactation. We hypothesize that adjunct aripiprazole will resolve hormonal effects in women with symptomatic hyperprolactinemia stabilized on risperidone (or paliperidone).
Time Frame: 16 Weeks
Population: 13 of the 20 Aripiprazole participants had lack of menstruation a the start of the study, and 11 of the 18 participants receiving placebo had lack of menstruation a the start of the study, therefore the analysis of return of menstruation is based on 24 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 13 | 11
Participants | 11 | 7

2. Secondary Outcome: To Test Whether Adjunctive Aripiprazole Will Improve Quality/Perceived Quality of Life.
Description: We will measure if patients' symptoms improve, improvement in their sexual dysfunction or distress and if they feel better with the elimination of the side effects. We hypothesize that aripiprazole will improve psychiatric symptoms, quality of life, sexual functioning and perceived wellness relative to placebo in women stabilized on risperidone (or paliperidone).
Time Frame: 16 Weeks
Population: 14 of the 20 participants receiving Aripiprazole and 11 of the 18 participants receiving placebo reported sexual dysfunction at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 14 | 11
Participants | 7 | 1

ADVERSE EVENTS:
Time Frame: Weekly for the 16 week study
Arm/Group | Aripiprazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 17/20 | 16/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=20) | Placebo (N=18)
Abdominal Pain (General disorders) | 7 | 6
Anorexia (Metabolism and nutrition disorders) | 4 | 4
Bruising Easily (General disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 6 | 5
Diarrhea (Gastrointestinal disorders) | 9 | 7
Dizziness (General disorders) | 5 | 4
Dry Mouth (General disorders) | 6 | 4
Euresis (General disorders) | 5 | 2
Fever (General disorders) | 1 | 2
Headache (General disorders) | 6 | 5
Insomnia (General disorders) | 8 | 3
Malaise (General disorders) | 7 | 5
Mucosal ulceration (General disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 10 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Restlessness (General disorders) | 5 | 2
Salavation (General disorders) | 4 | 5
Sedation (General disorders) | 7 | 6
Sore Throat (General disorders) | 2 | 4
Stiffness (Musculoskeletal and connective tissue disorders) | 5 | 5
Tinnitus (General disorders) | 7 | 2
Tremor (General disorders) | 8 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 10 | 7
Weight Loss (Metabolism and nutrition disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No